CLINICAL TRIAL: NCT00427752
Title: Diagnostic Transluminal Endoscopic Peritoneoscopy
Brief Title: Abdominal Exploration Without Incisions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jeffrey Hazey (Other)
Collaborators: Stryker Nordic (Industry); Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Hazey, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2006H0120
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Pancreatic Cancer
Keywords: Transgastric; Endoluminal; Peritoneoscopy; Diagnostic; Feasibility
MeSH Terms: conditions — Pancreatic Neoplasms; Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whipple (Experimental): Patients with pancreatic cancer who will proceed to a Whipple procedure.
  Interventions: Procedure: Transgastric endoscopic peritoneoscopy.

INTERVENTIONS:
Procedure: Transgastric endoscopic peritoneoscopy. — Exploration of the abdominal area

SUMMARY:
This study is being conducted to determine whether an endoscope, (a small, flexible tube with a camera mounted on the end) passed down through the throat, through the stomach, and into the abdomen can safely and accurately examine the organs and tissue of the abdomen and take biopsies if needed. We wish to determine if this endoscopic diagnostic route is as efficient as the laparoscopic diagnostic route, which is currently the standard of care.

DETAILED DESCRIPTION:
We propose to investigate the efficacy of transgastric endoscopic peritoneoscopy with endoscopic biopsy in patients undergoing diagnostic laparoscopy and who will require a concurrent gastrotomy for placement of a PEG, gastrojejunostomy or gastric resection.

We hypothesize that diagnostic endoscopic peritoneoscopy can be done safely with adequate visualization of the abdominal cavity to direct clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic Cancer undergoing staging laparoscopy
* Staging or diagnostic laparoscopy in anyone needing enteral access

Exclusion Criteria:

* Lack of consent
* Intra-abdominal adhesions precluding diagnostic laparoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
1) That transgastric endoscopic peritoneoscopy is feasible. | 4/12

SECONDARY OUTCOMES:
That bacterial abdominal contamination is not clinically significant. | 04/11

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Hazey, MD, Principal Investigator — Ohio State University; William S Melvin, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Center for Minimally Invasive Surgery, Columbus, Ohio, United States

REFERENCES:
- [Background] Narula VK, Hazey JW, Renton DB, Reavis KM, Paul CM, Hinshaw KE, Needleman BJ, Mikami DJ, Ellison EC, Melvin WS. Transgastric instrumentation and bacterial contamination of the peritoneal cavity. Surg Endosc. 2008 Mar;22(3):605-11. doi: 10.1007/s00464-007-9661-6. Epub 2007 Nov 20. PMID 18027034
- [Background] Cios TJ, Reavis KM, Renton DR, Hazey JW, Mikami DJ, Narula VK, Allemang MT, Davis SS, Melvin WS. Gastrotomy closure using bioabsorbable plugs in a canine model. Surg Endosc. 2008 Apr;22(4):961-6. doi: 10.1007/s00464-007-9530-3. Epub 2007 Aug 19. PMID 17710490
- [Background] Hazey JW, Dunkin BJ, Melvin WS. Changing attitudes toward endolumenal therapy. Surg Endosc. 2007 Mar;21(3):445-8. doi: 10.1007/s00464-006-9001-2. PMID 17054006
- [Background] Malik A, Mellinger JD, Hazey JW, Dunkin BJ, MacFadyen BV Jr. Endoluminal and transluminal surgery: current status and future possibilities. Surg Endosc. 2006 Aug;20(8):1179-92. doi: 10.1007/s00464-005-0711-7. Epub 2006 Jul 24. PMID 16865615
- [Result] Hazey JW, Narula VK, Renton DB, Reavis KM, Paul CM, Hinshaw KE, Muscarella P, Ellison EC, Melvin WS. Natural-orifice transgastric endoscopic peritoneoscopy in humans: Initial clinical trial. Surg Endosc. 2008 Jan;22(1):16-20. doi: 10.1007/s00464-007-9548-6. Epub 2007 Aug 14. PMID 17701250